

Page 1/31

## MIST 2

## STATISTICAL ANALYSIS PLAN

A clinical study to assess the feasibility of a controlled human *Plasmodium vivax* malaria infection model through experimental sporozoite infection in Thai adults.

Short title: MIST 2 study

Version 1.0

Date: 13 June 06 2022

| Written by: | |
|----------------------------------------|------|
| Prof. Mavuto Mukaka | |
| Print name & signature<br>Statistician | Date |
| Reviewed and approved by: | |
| Dr. Pongphaya Pongsuwan | |
| Print Name & signature | Date |
| Programme Manager | |

Template No.: T23-02 Effective Date: 27 May 2020

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022



| STATISTICAL ANALYSIS PLAN | |
|-----------------------------------------|----------|
| Assist. Prof. Borimas Hanboonkunupakarn | |
| Print Name & signature | <br>Date |
| Site Principal Investigator | |
| Dr. Wanlapa Roobsoong | |
| Print Name & signature | <br>Date |
| Investigator | |
| Dr. Sadudee Chotirat | |
| Print Name & signature | <br>Date |
| Researcher | |
| Dr. Wang Nguitragool | |
| Print Name & signature Researcher | Date |



| STATISTICAL ANALYSIS PLAN | |
|---------------------------------------------------|------|
| Prof. Jetsumon Sattabongkot Prachumsri | |
| Print Name & signature | Date |
| Co-Principal Investigator | |
| Prof. Nicholas Day | |
| Print Name & signature Co-Principal Investigator | Date |



# Contents

| 1. I | NTRODUCTION | 5 |
|---|---|---|
| 2. S | STUDY OBJECTIVES AND ENDPOINTS | 5 |
| 2.1 | Primary objective | 5 |
| 2.2 | Primary endpoint | 5 |
| 2.3 | Secondary objectives and endpoints | 6 |
| 3. S | STUDY DESIGN | 6 |
| 3.1 | General | 6 |
| 3.2 | Determination of sample size | 7 |
| 4. <i>A</i> | ANALYSIS | 7 |
| 4.1 | General considerations | 7 |
| | I.1.1 Data integrity | 8 |
| 4 | J.1.2 Data cleaning and verification | 8 |
| 4.2 | Dummy figure 1 – Study Profile | 9 |
| 4.3 | Study assessments | 10 |
| 4 | <b>1.3.1</b> Demographics and other baseline characteristics | 10 |
| 4 | 1.3.2 Clinical efficacy assessments (an example of a possible heading) | 12 |
| 4 | I.3.3 Pharmacokinetic assessments (an example of a possible heading) | 12 |
| 4 | 1.3.4 Adverse events | 12 |
| 4 | I.3.5 Cellular Response | 25 |
| 4 | I.3.6 Humoral Response | 28 |
| 4 | 1.3.7 Gametocyte Analysis | 31 |

### 1. INTRODUCTION

This project is the second part of a 5-year research program entitled "Malaria Infection Study in Thailand (MIST)" and known as MIST2. MIST2 primary objectives are to assess the safety and feasibility of blood-stage controlled human *P. vivax* malaria infection (CHMI) in healthy adult Thai volunteers through experimental injection of cryopreserved *P. vivax* infected erythrocytes, and to choose the optimal inoculation dose for future *P. vivax* CHMI studies. In this study, blood-stage CHMI will be conducted in 8 volunteers per inoculum stock who will be infected with *P. vivax* by experimental injection with cryopreserved *P. vivax* infected erythrocytes, which were collected in MIST1. As there are currently 2 stocks of inocula from 2 volunteers in the MIST1 study, which have different quantity and stage of parasites. The total number of volunteers would be up to 16. The volunteers will be monitored closely as inpatients in the Hospital for Tropical Diseases, and will be treated according to the Research Proposal Submission Form.

This documents sets out the statistical analysis plan for a MIST 2 to assess the feasibility and safety study and choosing the optimal inoculation dose for future *P. vivax* CHMI studies.

#### 2. STUDY OBJECTIVES AND ENDPOINTS

## 2.1 PRIMARY OBJECTIVE

- a) To assess the safety and feasibility of blood-stage controlled human *P. vivax* malaria infection in healthy adult Thai volunteers through experimental injection of cryopreserved *P. vivax* infected erythrocytes at different doses.
- b) To choose the optimal inoculation dose for future *P. vivax* CHMI studies.

### 2.2 PRIMARY ENDPOINT

a) Safety and feasibility of primary *P. vivax* blood-stage CHMI, as measured by (S)AE occurrences and successful infection (development of detectable persistent parasitaemia by thick blood film +/- clinical symptoms).

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 5/31



b) Choosing the optimal inoculation dose for future *P. vivax* CHMI studies, which will be the lowest concentration that produces a reliable infection within a comparable timeframe as compare to the highest concentration.

#### 2.3 SECONDARY OBJECTIVES AND ENDPOINTS

- a) To assess the immune response to *P. vivax* infection in volunteers, through experimental injection of *P. vivax* infected erythrocytes. The endpoint of this objective is immune response to experimental *P. vivax* infection through bloodstage challenge, as measured by antibody, cytokines, B cell and T cell responses.
- b) To assess gametocytaemia during *P. vivax* infection in volunteers, through experimental injection of *P. vivax* infected erythrocytes. The endpoint of this objective is gametocytaemia, as measured by qPCR in experimental *P. vivax* infection through blood-stage challenge.
- c) To assess transmission of gametocytes from infected volunteers to Anopheles mosquitoes. The endpoint of this objective is transmissibility of gametocytes from the infected volunteer to Anopheles mosquito vector.

### 3. STUDY DESIGN

## 3.1 GENERAL

This blood-stage *P. vivax* human challenge study conducted for the first time in Asia has two primary aims: (1) to assess the safety and feasibility of the challenge model using the bank of cryopreserved *P. vivax* infected erythrocyte inocula prepared during the MIST1 study, and (2) to determine the optimal inoculation dose for future *P. vivax* CHMI studies. This will be assessed by intravenously injecting the volunteers with four different doses of inoculum: whole dose and 1:5, 1:10, and 1:20 dilutions. If safe and feasible, this study will serve as the basis for a challenge model for future *P. vivax* candidate vaccine efficacy studies. The secondary objectives are to determine the immune response to *P. vivax* infection, the resulting gametocytaemia, and transmissibility of the gametocytes from the infected volunteers.

Healthy, Thai adults aged between 20 and 55 years will be recruited and randomized at the Faculty of Tropical Medicine, Mahidol University in Bangkok.

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 6/31



CHMI will be induced by injection of *P. vivax* infected erythrocytes and all follow-up in the post-challenge period will be performed at the Faculty of Tropical Medicine, Mahidol University in Bangkok.

Volunteers will have blood taken at regular intervals post-CHMI to assess the immune response to *P. vivax* infection, as well as parasite growth dynamics and gametocytaemia. We will also assess transmission of *P. vivax* gametocytes from the infected volunteers to mosquitos using a membrane feeding assay (MFA).

Close monitoring will continue until volunteers meet criteria for treatment or until 21 days after challenge, when treatment will be started empirically.

Therapy will be with a standard course of chloroquine where not contraindicated. As infection will be induced via intravenous injection of blood-stage parasites, there will be no liver-stage infection and no hypnozoite formation, thereby eliminating the need for radical cure with primaquine therapy. Follow-up at study site will be up to 1 year after antimalarial treatment initiated.

#### 3.2 DETERMINATION OF SAMPLE SIZE

In order to find the optimum dose of each blood-stage inoculum (the lowest concentration that the volunteers reliably develop infection, i.e., 2/2, within the comparable time frame as compare to the highest concentration and within 21 days), one blood-stage inoculum stock will be tested in 4 different doses: whole dose inoculum (neat vial), 1:5, 1:10, and 1:20 dilution. Each dose will be inoculated into two volunteers resulting in 8 volunteers. As two stocks of blood-stage inoculum were prepared from MIST1, 16 volunteers will be recruited: 8 to be challenged with inoculum stock 1, and 8 with inoculum stock 2.

#### 4. ANALYSIS

### 4.1 GENERAL CONSIDERATIONS

The feasibility and safety of blood-stage controlled human *P. vivax* malaria infection, will be declared if there will be a successful infection in at least one of the 8 volunteers



from each blood bank i.e. if there will be development of detectable persistent parasitaemia +/- clinical symptoms.

The success of this study will also be declared if infection is successful and we are able to choose the optimal inoculation dose for future *P. vivax* CHMI studies.

The safety of this challenge study will be assessed by summarising and evaluating the SAEs and the AEs regarding severity and relatedness to the challenge.

### **4.1.1** Data integrity

This study will be conducted in compliance with the protocol, relevant Standard Operating Procedures (SOPs), Work Instructions (WIs), Good Clinical Practice (GCP) and the applicable regulatory requirement(s). All the analyses will be performed on clean data only.

## **4.1.2** Data cleaning and verification

All data will be cleaned and verified prior to statistical analysis. The study site will be visited by the Monitor periodically at times agreed on with the Investigator. At the time of each monitoring visit, the Monitor will review the completed CRFs to ascertain that all items have been completed and that the data provided are accurate and obtained in the manner specified in the protocol. The Monitor will also check that the data in the CRF are consistent with the clinical records (Source Data Verification [SDV]) and that study results are recorded completely and correctly. Study Specific Audit will also be done to assess the clinical and laboratory study activities compliance with study protocol, SOPs and Plans, local QMS procedures, applicable standards and guidelines. The data manager will ensure that clean data is submitted to the statistician for analysis. The statistician will cross-check that the available data for analysis is clean. Any data cleaning queries will need to be resolved before statistical analyses.

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 8/31



#### 4.2 **DUMMY FIGURE 1 – STUDY PROFILE**



Page 9/31 Template No.: T23-02 Effective Date: 27 May 2020

## 4.3 STUDY ASSESSMENTS

## **4.3.1** Demographics and other baseline characteristics

The following baseline characteristics for each participant will be described and summarized for all participants in Table 1 below. Variables such as age, heart rate, respiratory rate, and laboratory data will be summarized using median and range. Continuous variables such as weight, height and hemoglobin will be summarized using mean and standard deviation. Categorical variables such as sex and symptoms will be summarized using frequencies. We will also compare the baseline characteristics for stock1 and stock2.

Table 1 Baseline Characteristics of the Subjects.

| Characteristics | Neat vial | Dose 1:5 | Dose 1:10 | Dose 1:20 | Total |
|---|---|---|---|---|---|
| Age (years), mean (IQR) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Male, n (%) | x (%) | x (%) | x (%) | x (%) | x (%) |
| Body temperature (°C), median (IQR) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Blood pressure (mmHg), | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| (Systolic/Diastolic), median (IQR) | | | | | |
| Heart rate (beats/min), median (IQR) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Respiratory rate (breaths/min), | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| median (IQR) | | | | | |
| Weight (kg), median (IQR) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Height (cm), median (IQR) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Haematology | | | | | |
| WBC (103/μL), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| RBC (10 <sup>6</sup> /μL), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Haemoglobin (g/dL), mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Haematocrit (%),median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Pletelets (103/μL), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Neutrophil (%),median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Lymphocyte (%),median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 10/31



| Characteristics | Neat vial | Dose 1:5 | Dose 1:10 | Dose 1:20 | Total |
|---|---|---|---|---|---|
| Monocyte (%),median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Eosinophil (%), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Basophil (%),median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Other abnormal WBC, median | yay (yay) | , (vo.) | vov (vov) | vov (vov) | vov (vov) |
| (IQR) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Platelet smear, n(%) | | | | | |
| Adequate | x (%) | x (%) | x (%) | x (%) | x (%) |
| Decrease | x (%) | x (%) | x (%) | x (%) | x (%) |
| Increase | x (%) | x (%) | x (%) | x (%) | x (%) |
| Biochemistry | | | | | |
| FBS (mg/dL), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| BUN (mg/dL), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Creatinine (mg/dL), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Total bilirubin (mg/dL), median | , n, (, n, , , n, ) | | .a.(.aa.) | .a. (.aa.) | () |
| (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| eGFR (mL/min), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Alkaline Phosphatase (U/L), | , , | , , | , , | , , | , , |
| median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| AST (U/L), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| ALT (U/L), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Albumin (g/dL), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Globulin (U/L), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Sodium (mmol/L), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Potassium (mmol/L), median | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| (IQR) | | | | | |
| Calcium (mg/dL), median (IQR) | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| Magnesium (mg/dL), median | xx (xx - xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| (IQR) | | | | | |
| Chloride (mmol/L), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 11/31



| Characteristics | Neat vial | Dose 1:5 | Dose 1:10 | Dose 1:20 | Total |
|---|---|---|---|---|---|
| Bicarbonate (mmol/L), median (IQR) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |
| etc | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) | xx (xx – xx) |

## **4.3.2** Clinical efficacy assessments (an example of a possible heading)

No clinical efficacy planned for MIST 2. However, Optimal dose will be assessed.

Referring from the protocol the optimal inoculation dose for future P. vivax CHMI studies is the lowest concentration that produces a reliable infection within a comparable timeframe as compared to the highest concentration.

## **4.3.3** Pharmacokinetic assessments (an example of a possible heading)

No PK analyses planed for MIST 2

#### **4.3.4** Adverse events

Adverse events will be summarized as shown in Tables 2a, 2b, 3a and 3b below. Firstly, all events will be captured.ie. including multiple events in an individual. Thereafter the number of individuals with at least an event will be recorded and the highest grade will be presented.

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 12/31 Effective Date: 27 May 2020



# Table 2a Adverse events during the admission phase before treatment as assessed by blood-stage stock

| | Stock1 blood- | stock2 blood- | Total |
|----------------------------------|---------------|---------------|-----------|
| Adverse event | stage (n=xx) | stage (n=xx) | (n=xx) |
| CTCAE Grade 1 or 2 of symptom or | | | |
| disease, x/n (%) | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| CTCAE Grade 1 or 2 abnormal | | | |
| laboratory findings, x/n (%) | | | |
| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Alanyl transfarase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Aspartate transfarase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 13/31



| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) |
|----------------------------------|-----------|-----------|-----------|
| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| CTCAE Grade 3 or 4 of symptom or | | | |
| disease, x/n (%) | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Other* | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| CTCAE Grade 3 or 4 abnormal | | | |
| laboratory findings, x/n (%) | | | |
| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Alanyl transferase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Aspartate transferase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 14/31



| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) |
|--------------|-----------|-----------|-----------|
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) |

<sup>\*</sup>Other symptoms or signs

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 15/31



# Table 2b Adverse events during the admission phase before treatment as assessed by dose.

| | Total | Neat vial | Dose 1:5 | Dose | Dose | P-value |
|---|---|---|---|---|---|---|
| Adverse event | event | | | 1:10 | 1:10 | |
| | (n=xx) | (n=xx) | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| CTCAE Grade 1 or 2 of symptom or | | | | | | |
| disease, x/n (%) | | | | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| CTCAE Grade 1 or 2 abnormal | | | | | | |
| laboratory findings, x/n (%) | | | | | | |
| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alanyl transfarase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Aspartate transfarase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 16/31



| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
|---|---|---|---|---|---|---|
| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| CTCAE Grade 3 or 4 of symptom or | | | | | | |
| disease, x/n (%) | | | | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Other* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| CTCAE Grade 3 or 4 abnormal | | | | | | |
| laboratory findings, x/n (%) | | | | | | |
| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alanyl transferase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Aspartate transferase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 17/31



| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
|---|---|---|---|---|---|---|
| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |

<sup>\*</sup>Other symptoms or signs

Table 3a Adverse events during the treatment phase as assessed by blood-stage stock.

| | Stock1 blood- | stock2 blood- | Total |
|---|---|---|---|
| Adverse event | stage | stage | |
| | (n=xx) | (n=xx) | (n=xx) |
| CTCAE Grade 1 or 2 of symptom or disease, | | | |
| x/n (%) | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| CTCAE Grade 1 or 2 abnormal laboratory | | | |
| findings, x/n (%) | | | |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 18/31

# MORU: Tropical Health Network

# STATISTICAL ANALYSIS PLAN

| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) |
|---|---|---|---|
| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Alanyl transfarase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Aspartate transfarase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| CTCAE Grade 3 or 4 of symptom or disease, | | | |
| x/n (%) | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| CTCAE Grade 3 or 4 abnormal laboratory | | | |
| findings, x/n (%) | | | |
| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) |



| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
|-----------------------------|-----------|-----------|-----------|
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Alanyl transfarase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Aspartate transfarase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) |

<sup>\*</sup>Other symptoms or signs

# Table 3b Adverse events during the treatment phase as assessed by dose.

| Adverse event | Total event (n=xx) | Neat vial | Dose 1:5<br>(n=xx) | Dose<br>1:10<br>(n=xx) | Dose<br>1:10<br>(n=xx) | P-value<br>(n=xx) |
|---|---|---|---|---|---|---|
| CTCAE Grade 1 or 2 of symptom or disease, x/n (%) | | | | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 20/31

# MORU: Tropical Health Network

# STATISTICAL ANALYSIS PLAN

| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
|---|---|---|---|---|---|---|
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| CTCAE Grade 1 or 2 abnormal | | | | | | |
| laboratory findings, x/n (%) | | | | | | |
| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alanyl transfarase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Aspartate transfarase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| CTCAE Grade 3 or 4 of symptom | | | | | | |
| or disease, x/n (%) | | | | | | |
| Fever | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Headache | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Myalgia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Palpitation | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Dizziness | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Chills | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Abdominal pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Profuse sweating | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Anorexia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Nausea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Vomitting | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Diarrhea | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Muscle pain | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Anemia | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |



| Other* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
|---|---|---|---|---|---|---|
| CTCAE Grade 3 or 4 abnormal | | | | | | |
| laboratory findings, x/n (%) | | | | | | |
| Creatinine | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Total bilirubin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alkaline phosphatase | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Alanyl transfarase (ALT) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Aspartate transfarase (AST) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Nadir Haemoglobin | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| WBC | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Platelet | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |
| Other signs* | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | xx/xx (%) | 0.xxx |

<sup>\*</sup>Other symptoms or signs

Relationship of adverse events to either treatment or infection will be summarized in Table 4 below.

Table 4 Distribution of adverse events by relationship to study procedures.

| During admission | (infection) phase | During treatment phase | |
|---|---|---|---|
| | Possibly, | | Possibly, |
| Any relationship | probably, | Any relationship | probably, |
| to study drugs | definitely related | to study drugs | definitely related |
| (n=xx) | to study drugs | (n=xx) | to study drugs |
| | (n=xx) | | (n=xx) |
| x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| | Any relationship to study drugs (n=xx) x/xx (x.x) x/xx (x.x) x/xx (x.x) x/xx (x.x) x/xx (x.x) x/xx (x.x) | Any relationship to study drugs (n=xx) definitely related to study drugs (n=xx) x/xx (x.x) x/xx (x.x) | Possibly, Any relationship to study drugs to study drugs (n=xx) (n=xx) |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 22/31



| Diarrhea | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
|---|---|---|---|---|
| Dizziness | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Dry mouth | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Dyspepsia | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Fatigue | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Fever | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Flushing | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Gingivitis | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Headache | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Insomnia | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Malaise | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Maculopapular | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Mucositis oral | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Myalgia | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Nausea | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Neck pain | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Palpitation | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Profuse sweating on palms & soles | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Pruritus. | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Sore throat | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Tachycardia | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Urinary tract infection | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Urticaria | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Vomiting | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Other signs* | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |

Values in cells are x/n (%).

Serious adverse events will be summarized in Tables 5a and 5b below.

<sup>\*</sup>Other symptoms or signs



# Table 5a Serious adverse events as assessed by dose.

| Serious adverse event | Total event (n=xx) | Neat vial | Dose 1:5<br>(n=xx) | Dose<br>1:10<br>(n=xx) | Dose<br>1:10<br>(n=xx) | P-value<br>(n=xx) |
|---|---|---|---|---|---|---|
| Death, x/n (%) | xx/xx (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | 0.xxx |
| Life-threatening event, x/n (%) | xx/xx (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | 0.xxx |
| Persistent or significant disability or incapacity, x/n (%) | xx/xx (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | 0.xxx |
| Transfer of inpatient care to the intensive care unit, x/n (%) | xx/xx (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | 0.xxx |
| An important medical event, x/n (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | 0.xxx |
| Congenital anomaly or birth defect, x/n (%) | xx/xx (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | 0.xxx |

# Table 5b Serious adverse events by relationship to study procedures.

| | During admiss | | During treatment phase | |
|---|---|---|---|---|
| Adverse event | Any relationship to study drugs (n=xx) | Possibly, probably, definitely related to study drugs (n=xx) | Any relationship to study drugs (n=xx) | Possibly, probably, definitely related to study drugs (n=xx) |
| Death, x/n (%) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Life-threatening event, x/n (%) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| Persistent or significant disability or incapaci-ty, x/n (%) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 24/31



| | During admiss | | During treatment phase | |
|---|---|---|---|---|
| Adverse event | Any relationship to study drugs (n=xx) | Possibly, probably, definitely related to study drugs (n=xx) | Any relationship to study drugs (n=xx) | Possibly, probably, definitely related to study drugs (n=xx) |
| Transfer of inpatient care to the intensive care unit, x/n (%) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |
| An important medical event, x/n (%) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) | x/xx (x.x) |

A detailed listing will also be shown.

## <u>Immune response</u>

The assessment of the immune response to *P. vivax* infection in volunteers, through experimental injection of *P. vivax* infected erythrocytes will be analysed as detailed below:

## **4.3.5** Cellular Response

The dynamic of cellular response will be determined using peripheral blood mononuclear cells (PBMCs). The data will be summarized as frequencies, percentages (%), and expression level (median fluorescence intensity (MFI)) as shown in Table 6 below. A spaghetti plot will be constructed and presented to show the profile of each of the important parameters over time across the participants. The profiles will also be presented as a plot of box and whisker plot indicating the profile of median and quartiles of the absolute parameters over-time. Where tests of hypothesis will be necessary, paired tests such as Wilcoxon's signed rank test will be used to compare parameters at a specified day with the baseline will be performed. Caution will be considered when interpreting such significant tests considering that sample sizes are very small. Tests of significance will be performed at 5% significance level. Stata software of at least version 15.0 will be used to analyse the data and make plots. Some plots will be done in GraphPad Prism where necessary. MFI value will be analysed and plotted by FlowJo software.

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 25/31



# Table 6 Immunological profile (frequency, %, MFI)

| Immune cell<br>subset | Screening phase<br>(Baseline) | | Admission phase | | | Follow-up phase | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Within 14<br>days prior<br>to Day 0 | Admission<br>Day-1 | Day <sub>4</sub> | Day<br>qPCR <sup>+</sup> | Day <sub>reach</sub> treatment criteria | Day <sub>Rx7</sub> | Day <sub>Rx28</sub> | Day <sub>Rx60</sub> | Day <sub>Rx90</sub> | Day <sub>Rx180</sub> | Day <sub>Rx1</sub> year |
| Conventional | | | | | | | | | | | |
| Dendritic cell | | | | | | | | | | | |
| (cDC) | | | | | | | | | | | |
| Myeloid | | | | | | | | | | | |
| Dendritic cell | | | | | | | | | | | |
| (MDC) | | | | | | | | | | | |
| Plasmacytoid | | | | | | | | | | | |
| Dendritic cell | | | | | | | | | | | |
| (PDC) | | | | | | | | | | | |
| Natural Killer | | | | | | | | | | | |
| (NK) | | | | | | | | | | | |
| Natural Killer T<br>(NKT) | | | | | | | | | | | |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 26/31



| Immune cell | Screening phase<br>(Baseline) | | Adı | Admission phase | | | Follow-up phase | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| subset | Within 14<br>days prior<br>to Day 0 | Admission<br>Day-1 | Day <sub>4</sub> | Day<br>qPCR <sup>+</sup> | Day <sub>reach</sub> treatment criteria | Day <sub>Rx7</sub> | Day <sub>Rx28</sub> | Day <sub>Rx60</sub> | Day <sub>Rx90</sub> | Day <sub>Rx180</sub> | Day <sub>Rx1Year</sub> |
| Mucosal Associated Invariant T cell (MAIT) | | | | | | | | | | | |
| Helper T-cell Cytotoxic T-cell Regulatory T-cell γδ T-cell | | | | | | | | | | | |
| Typical B-cell Plasmablast | | | | | | | | | | | |



## **4.3.6** Humoral Response

## Cytokine response (median fluorescence intensity, relative antibody unit)

The level of cytokine responses related blood stage inoculum will be assessed by using Multiplex Bead Based Immunoassay (Luminex) and/or ELISA, and summarised in Table 7 below. Luminex and/or ELISA will be used to explore the level of antibodies and cytokines responses during different phases of infection. P-values for the test of significance will be indicated where applicable. However, Caution will be considered when interpreting such significant tests considering that sample sizes are very small.

Table 7 Cytokine/Chemokine response profile (plasma level pg/ml)

| Cytokine/<br>Chemokine | Screening phase<br>(Baseline) | | Ad | Admission phase | | | Follow-up phase | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Within 14<br>days prior<br>to Day 0 | Admission<br>Day-1 | Day <sub>4</sub> | Day<br>qPCR <sup>+</sup> | Day <sub>reach</sub> treatment criteria | Day <sub>Rx7</sub> | Day <sub>Rx28</sub> | Day <sub>Rx60</sub> | Day <sub>Rx90</sub> | Day <sub>Rx180</sub> | Day <sub>Rx1Year</sub> |
| FGF basic | | | | | | | | | | | |
| Eotaxin | | | | | | | | | | | |
| G-CSF | | | | | | | | | | | |
| GM-CSF | | | | | | | | | | | |
| IFN-γ | | | | | | | | | | | |
| IL-1β | | | | | | | | | | | |

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 28/31



| Cytokine/<br>Chemokine | | ng phase<br>eline) | Admission phase | | | Follow-up phase | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Within 14<br>days prior<br>to Day 0 | Admission<br>Day-1 | Day₄ | Day<br>qPCR <sup>+</sup> | Day <sub>reach</sub> treatment criteria | Day <sub>Rx7</sub> | Day <sub>Rx28</sub> | Day <sub>Rx60</sub> | Day <sub>Rx90</sub> | Day <sub>Rx180</sub> | Day <sub>Rx1Year</sub> |
| IL-1ra | | | | | | | | | | | |
| IL-2 | | | | | | | | | | | |
| IL-4 | | | | | | | | | | | |
| IL-5 | | | | | | | | | | | |
| IL-6 | | | | | | | | | | | |
| IL-7 | | | | | | | | | | | |
| IL-8 | | | | | | | | | | | |
| IL-9 | | | | | | | | | | | |
| IL-10 | | | | | | | | | | | |
| IL-12 (p70) | | | | | | | | | | | |
| IL-13 | | | | | | | | | | | |
| IL-15 | | | | | | | | | | | |



| Ortokino | | ng phase<br>eline) | Admission phase | | | Follow-up phase | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cytokine/<br>Chemokine | Within 14<br>days prior<br>to Day 0 | Admission<br>Day-1 | Day <sub>4</sub> | Day<br>qPCR <sup>+</sup> | Day <sub>reach</sub> treatment criteria | Day <sub>Rx7</sub> | Day <sub>Rx28</sub> | Day <sub>Rx60</sub> | Day <sub>Rx90</sub> | Day <sub>Rx180</sub> | Day <sub>Rx1Year</sub> |
| IL-17A | | | | | | | | | | | |
| IP-10 | | | | | | | | | | | |
| MCP-1 (MCAF) | | | | | | | | | | | |
| MIP-1α | | | | | | | | | | | |
| МΙР-1β | | | | | | | | | | | |
| PDGF-BB | | | | | | | | | | | |
| RANTES | | | | | | | | | | | |
| TNF-α | | | | | | | | | | | |
| VEGF | | | | | | | | | | | |
| TGF-β1 | | | | | | | | | | | |



## **4.3.7** *Gametocyte Analysis*

Another secondary objective of MIST2 study is to assess gametocytaemia following *P. vivax* infection delivered by blood-stage inoculum. The endpoint is gametocytaemia pretreatment, as measured by qRT-PCR.

The endpoint for gametocyte detection will be the Pvs25 gene transcript copy number/ul blood collected at each time point as follows: challenge day; day 1 to 5 or up to day of treatment and during subsequent days of follow-up. The data will be summarized using the geometric mean and standard deviation/error at each time point. The trend in geometric means will be assessed and where necessary will be presented graphically using trend lines.

Study code: MIST 2 .Edit check List version: 1.0 Date: 13062022 Page 31/31